CLINICAL TRIAL: NCT03538353
Title: Patients' Perspectives About a Pain Education Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Erin Dannecker, Assoc Prof & Director of Scholarly Activity - Physical Therapy, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSIRB# 2010486
Record Dates: First submitted 2018-04-30; First posted 2018-05-29 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Education Video (Other): Participants will watch a pain education video and then answer several questions.
  Interventions: Other: pain education video

INTERVENTIONS:
Other: pain education video — The video was made for the DOD and VHA to educate their soldiers and veterans about chronic pain.

SUMMARY:
The overall goal of this single session semi-structured interview project is to explore the validation and contradiction of the preexisting pain beliefs in patients with chronic pain.

Aim 1: After patients watch an educational video, explore occurrences of perceived validation and contradiction and the impact of validation and contradiction on pain beliefs, emotion, and pain.

Aim 2: Obtain patients' recommendations for improving the educational value of the video.

DETAILED DESCRIPTION:
The long-term goal is to reduce disability in patients with chronic pain by improving communication about pain among patients, caregivers, and health care providers (HCPs). The proposed study addresses the long-term goal by conducting a project that investigates the validation and contradiction of patients' preexisting pain beliefs during pain education. Completion of the proposed project will advance the literature on validation and contradiction in patients with chronic pain by (1) focusing on a pain education resource instead of dyadic communication, (2) modifying a measure of validation and contradiction for relevance to an education resource, (3) exploring erroneous perceptions of validation and contradiction, (4) examining the impact of validation and contradiction on pain beliefs, and (5) obtaining patients' recommendations for a popular pain education film. The information gained will be used to improve pain education resources to increase their beneficial effects on pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older;
* new patient of the CPMC;
* living independently; and
* self-reported recurrent or persistent pain on most days of the last year.

Exclusion Criteria:

* previously viewed the pain education video used in this project;
* insufficient hearing to communicate with an interviewer; and
* an inability to complete the session within the time allowable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
agreement and disagreement with preexisting beliefs | 1 day
  qualitatively assessed via thematic analysis of semi-structured interviews

SECONDARY OUTCOMES:
emotional response to agreement and disagreement with preexisting beliefs | 1 day
  qualitatively assessed via thematic analysis of semi-structured interviews
pain beliefs | 1 day
  qualitatively assessed via thematic analysis of semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Erin A Dannecker, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri - Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No